CLINICAL TRIAL: NCT05472727
Title: Comparison of Physical Fitness, Walking Speed, Reaction Time In Older Adults With and Without Mild Cognitive Impairment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Zeynep SAG, PT, Dokuz Eylul University
Other Study IDs: 6987-GOA
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Reaction Time; Physical Fitness
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group (mild cognitive impairment): geriatric population with mild cognitive impairment
  Interventions: Other: reaction time test; Other: Physical fitness test
- Control Group (healthy elderly): healthy older adults without cognitive impairment
  Interventions: Other: reaction time test; Other: Physical fitness test

INTERVENTIONS:
Other: reaction time test — Reaction time tests consist of 3 sub-parameters as simple reaction time, selective reaction time and distinctive reaction time. Participants will do these tests on the computer.
Other: Physical fitness test — The physical fitness test will be evaluated with the senior fitness test used for geriatrics and the 8 meter walking speed test.

SUMMARY:
The aim of the study is to compare physical fitness, walking speed and hand reaction time measurements in older adults with different cognition levels according to the Montreal Cognitive Assessment Scale (MOCA).

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Volunteering to participate in the study
* 10 meters independent walking
* Being diagnosed with mild cognitive dysfunction
* Not being diagnosed with cognitive dysfunction
* Having received five years of basic education

Exclusion Criteria:

* Having had an upper or lower extremity surgery in the last 6 months
* Having a health problem that prevents completing the tests in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: elderly people who are healthy or with mild cognitive impairment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
reaction time | Participants are expected to complete the 3 sub-parameters of reaction time measurements in an average of 20 minutes, including rest periods
  reaction time

SECONDARY OUTCOMES:
physical fitness | Physical fitness tests are expected to take an average of 20 minutes.
  physical capacity of the person

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Engin Simsek, professor, Study Chair — iengin.simsek@gmail.com